CLINICAL TRIAL: NCT05829252
Title: Testing the Feasibility of a Novel Growth Monitoring Smartphone App
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 286683
Record Dates: First submitted 2023-03-06; First posted 2023-04-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Short Stature; Growth Disorders
Keywords: Height measurement; Child height; Short stature; Smartphone App; Digital Health
MeSH Terms: conditions — Dwarfism; Growth Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical trial is to test the acceptability, feasibility, accuracy and precision of the 'GrowthMonitor' smartphone app in a pilot population.

DETAILED DESCRIPTION:
The GrowthMonitor app will calculate height data using smartphone images of children taken by parents or carers in the home at two or more set time points. The app will convert height data from the image to a numerical height measurement in centimeters and this will be transferred to a central database hosted on a secure UK based server with additional relevant demographic data (gender, ethnicity, weight, date of birth, and parents' height).

The height and demographic data are transferred with an anonymous identifier to a GDPR-approved secure database on a UK based server. Critically, patient images and children's names will not be transferred, and only authorized users will have access to the data stored within the secure database.

The app will display a virtual growth chart providing the patient with a digital history of the child's growth over time. BMI will also be calculated and plotted on an age- and gender-appropriate chart. Ultimately, users of the app will need to create an account using a username (email address) and password. We will use their email address so that password resets can be sent along with reminders or alerts about their account.

Child's height in relation to his/her parental heights as well as longitudinal growth data will be analyzed within the secure UK based web server using existing growth monitoring algorithms.

1. Height compared to population-based height references (HSDS)
2. Distance from target height (calculated from parental heights, THSDSDEV)
3. HSDS change over time (ΔHSDS) -when more than one height measurement is available (taken >6 months apart)

Recorded heights will be compared with pre-established cut-off standards that define normal growth in an appropriate population. We envisage being able to incorporate ethnicity-matched reference population data as the app evolves. An automated outcome will be returned to the parent/carer, via in app notification or email, and will offer advice, for example, confirming normal growth or recommending appropriate medical contact.

Data will be stored in such a way that users can sync their old growth measurements on to any new / replacement smartphone handset and also 'sync' any measurements taken offline.

An accurate standing height measurement will be obtained using a calibrated stadiometer during a patient clinic visit. This 'gold standard' height measurement will be performed by a trained member of the research team and documented. This will be used to compare with the height obtained by the growth monitoring app in the clinic and subsequently at home.

ELIGIBILITY:
Inclusion Criteria:

* Children and young people (male and female) aged 1-18 yr receiving height measurements as part of their routine / prearranged attendance to a paediatric endocrinology or other paediatric out-patient appointment at Barts Health Trust.
* Participants require a smartphone to take part in the study.

Exclusion Criteria:

* Children under the age of 1 years
* Young people aged 16-18yr who lack capacity to consent
* Other individuals unable to reliably stand for an accurate height measurement e.g.

individuals with severe disability and/or confined to a wheelchair

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients attending prearranged new and follow-up outpatient appointments at the Children's Hospital at Barts Health Trust, London. Participants will be recruited through convenience sampling in order to maximize recruitment efforts during the time of the study. Data on gender, age, and height will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Reliability | At baseline
  Inter- and intra-rater reproducibility of the GrowthMonitor app
Agreement | At baseline
  Agreement between the GrowthMonitor app and wall-fixed stadiometer

SECONDARY OUTCOMES:
Usability | At 1 week
  Participants rate the usability of the GrowthMonitor app on a multiple-question 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Helen Storr, PhD, Principal Investigator — Queen Mary University, London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No